CLINICAL TRIAL: NCT00969202
Title: Phase 1 Study of Stereotactic Hypofractionated Radiosurgery of Low Grade Prostate Cancer/Early Stage
Brief Title: Stereotactic Hypofractionated Radiosurgery for Early Stage Prostate Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Diego Radiosurgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDRS0001
Record Dates: First submitted 2009-08-28; First posted 2009-09-01 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Cancer of the Prostate; Prostate Tumor; Novalis Tx; Novalis; Stereotactic Radiosurgery; Radiosurgery; Radiation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic Radiosurgery using NovalisTx (Experimental): Single arm study using the Novalis Tx to perform radiosurgery to treat low grade prostate cancer.
  Interventions: Radiation: Stereotactic Radiosurgery using the Novalis Tx

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery using the Novalis Tx — Five treatments given every other day.
  Other Names: Novalis Tx; Novalis

SUMMARY:
The purpose of this trial is to evaluate a short course of very focused (stereotactic) external beam radiation therapy for the treatment of early stage prostate cancer.

The investigators will gather scientific information about the tolerance and side effects this type of radiation. The investigators will then compare these results with those of standard 8 week course of external beam radiation therapy to see if this study treatment is equally or more effective in treating prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Gleason score ≤ 6 and low volume Gleason 7 (3+4)
* PSA < 10
* Clinical Stage of T2a or less
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior radiation treatment for prostate cancer
* Gleason score > 7
* PSA > 10
* Clinical Stage of T2b or greater

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
PSA decline measured through laboratory testing. | One month following radiosurgery through 5 year follow up

SECONDARY OUTCOMES:
Quality of life in relation to urinary, bowel and sexual function. Measured through a questionnaire at each follow up visit. | One month following radiosurgery through 5 years follow up.

CONTACTS AND LOCATIONS:
Overall Officials: P. Brian Volpp, MD, MPH, Principal Investigator — San Diego Radiosurgery/X-Ray Medical Group-Radiation Oncology
Locations (1):
- San Diego Radiosurgery at Palomar Medical Center, Escondido, California, United States